CLINICAL TRIAL: NCT06046105
Title: Efficacy of Adding Dexmedetomidine Versus Ibuprofen as an Adjuvant to Intraperitoneal Bupivacaine for Pain Control After Laparoscopic Gynecological Procedures: a Double-blind Randomized Comparative Study
Brief Title: Efficacy of Adding Dexmedetomidine Versus Ibuprofen as an Adjuvant to Intraperitoneal Bupivacaine for Pain Control After Laparoscopic Gynecological Procedures
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Wael El GHARABAWY, Assistant professor of anesthesiology, ICU, pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU R131/2023
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Pain, Acute
Keywords: dexmedetomidine, ibuprofen, bupivacaine, intraperitoneal, gynecological, laparoscopic, analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Randomized controlled comparative prospective clinical trial
Who Masked: Participant, Care Provider
Masking Description: The study drugs will be prepared in a ready-to-inject form by a separate anesthesiologist who is not involved in the study.
  This way, neither the patient nor the anesthesiologist administering the drug will be aware of the type of medication being used.
  The physician who will gather patient data is also unaware of the medications administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Bupivacaine group (Group B) (control group) (Sham Comparator): Patients will receive 50 ml of Bupivacaine 0.25% (125mg) diluted in 100 ml of normal saline. The drug will be injected intraperitoneally through trocars at the end of the surgery.
  Interventions: Drug: Administering intraperitoneal bupivacaine for pain control after laparoscopic gynecological procedures
- Bupivacaine/Ibuprofen group (Group BI) (Experimental): Patients will receive 50 ml of Bupivacaine 0.25% (125 mg) + 400 mg Ibuprofen diluted in 100 ml normal saline. The drug will be injected intraperitoneally through trocars at the end of the surgery.
  Interventions: Drug: Administering intraperitoneal bupivacaine plus Ibuprofen for pain control after laparoscopic gynecological procedures
- Bupivacaine/Dexmedetomidine group (Group BD): (Active Comparator): Patients will receive 20 ml of bupivacaine 0.25% (125 mg) + 1 µq/kg dexmedetomidine diluted in 100 ml normal saline. The drug will be injected intraperitoneally through trocars at the end of the surgery.
  Interventions: Drug: Administering intraperitoneal bupivacaine plus Dexmedetomidine for pain control after laparoscopic gynecological procedures

INTERVENTIONS:
Drug: Administering intraperitoneal bupivacaine for pain control after laparoscopic gynecological procedures — All patients will receive a standardized general anesthetic. Intravenous induction will be achieved with propofol, fentanyl (up to 2 µg/kg), rocuronium 0.6 mg/kg, and ondansetron 4 mg.
  Anesthesia will be maintained with 50% oxygen/ air mixture and isoflurane, intravenous fentanyl boluses (up to 3 µg/kg), rocuronium to maintain muscle relaxation, and intravenous fluids administered as Ringer's lactate (minimum of 20 mL/kg).
  All incision sites were infiltrated with 0.25% bupivacaine, and CO2 insufflation pressure was limited to a maximum of 15 mmHg.
  At the end of the procedure bupivacaine injection will be given by the surgeon through trocars intraperitoneally.
  Patients will be transferred to the post-anesthetic care unit (PACU) and the Modified Aldrete Score will be assessed and discharged after fulfilling an Aldrete score of ≥9.
  During the first 24 hr. after surgery, all patients will receive 1 gm paracetamol i.v. every 8 hr.
  Arms: Bupivacaine group (Group B) (control group)
Drug: Administering intraperitoneal bupivacaine plus Dexmedetomidine for pain control after laparoscopic gynecological procedures — All patients will receive a standardized general anesthetic. Intravenous induction will be achieved with propofol, fentanyl (up to 2 µg/kg), rocuronium 0.6 mg/kg, and ondansetron 4 mg.
  Anesthesia will be maintained with 50% oxygen/ air mixture and isoflurane, intravenous fentanyl boluses (up to 3 µg/kg), rocuronium to maintain muscle relaxation, and intravenous fluids administered as Ringer's lactate (minimum of 20 mL/kg).
  All incision sites were infiltrated with 0.25% bupivacaine, and CO2 insufflation pressure was limited to a maximum of 15 mmHg.
  At the end of the procedure bupivacaine plus Dexmedetomidine injection will be given by the surgeon through trocars intraperitoneally.
  Patients will be transferred to the post-anesthetic care unit (PACU) and the Modified Aldrete Score will be assessed and discharged after fulfilling an Aldrete score of ≥9.
  During the first 24 hr. after surgery, all patients will receive 1 gm paracetamol i.v. every 8 hr.
  Arms: Bupivacaine/Dexmedetomidine group (Group BD):
Drug: Administering intraperitoneal bupivacaine plus Ibuprofen for pain control after laparoscopic gynecological procedures — All patients will receive a standardized general anesthetic. Intravenous induction will be achieved with propofol, fentanyl (up to 2 µg/kg), rocuronium 0.6 mg/kg, and ondansetron 4 mg.
  Anesthesia will be maintained with 50% oxygen/ air mixture and isoflurane, intravenous fentanyl boluses (up to 3 µg/kg), rocuronium to maintain muscle relaxation, and intravenous fluids administered as Ringer's lactate (minimum of 20 mL/kg).
  All incision sites were infiltrated with 0.25% bupivacaine, and CO2 insufflation pressure was limited to a maximum of 15 mmHg.
  At the end of the procedure bupivacaine plus Ibuprofen injection will be given by the surgeon through trocars intraperitoneally.
  Patients will be transferred to the post-anesthetic care unit (PACU) and the Modified Aldrete Score will be assessed and discharged after fulfilling an Aldrete score of ≥9.
  During the first 24 hr. after surgery, all patients will receive 1 gm paracetamol i.v. every 8 hr.
  Arms: Bupivacaine/Ibuprofen group (Group BI)

SUMMARY:
The goal of this clinical trial is to compare the analgesic efficacy of adding dexmedetomidine versus ibuprofen to bupivacaine for intraperitoneal instillation after laparoscopic gynecological procedures. The main questions to answer are:

* Which is more effective for controlling postoperative pain within the first 24 hours after the procedure?
* Which is more convenient for the patients with fewer side effects and opioid consumption?

Participants will be asked to assess

* The postoperative pain severity by VAS score
* The onset of the first analgesic request
* The incidence of side effects like nausea and vomiting Researchers will compare the dexmedetomidine group, the ibuprofen group, and the bupivacaine (control) group to see which one will be superior to the others.

DETAILED DESCRIPTION:
The patients will be randomly allocated by simple randomization using a computer program into two equal groups by closed envelope technique:

Group 1: Bupivacaine/Ibuprofen group (BI): Patients will receive 50ml bupivacaine 0.25% (125 mg) + 400 mg Ibuprofen diluted in 100 ml normal saline.

Group 2: Bupivacaine/Dexmedetomidine group (BD): Patients will receive 20 ml bupivacaine 0.25% (125 mg) + 1 µq/kg dexmedetomidine diluted in 100 ml normal saline.

Group 3: Control group/Bupivacaine group (B): Patients will receive 50 ml Bupivacaine 0.25% (125mg) diluted in 100 ml normal saline.

All the previous drugs will be injected intraperitoneally through trocars at the end of the surgery.

All patients will be assessed preoperatively by careful history taking, full physical examination, laboratory evaluation, and other appropriate investigations.

At the preoperative visit, all patients will be instructed on how to evaluate their pain by using the visual analog scale (VAS) (range from 0-10., 0 =no pain, 10 = worst pain).

* Intraoperative settings:

All patients will receive a standardized general anesthetic. Intravenous induction will be achieved with propofol, fentanyl (up to 2 µg/kg), rocuronium 0.6 mg/kg, and ondansetron 4 mg. All patients will be intubated with an endotracheal tube and mechanically ventilated to maintain normocarbia. Anesthesia will be maintained with 50% oxygen/ air mixture and isoflurane, intravenous fentanyl boluses (up to 3 µg/kg), rocuronium to maintain muscle relaxation and intravenous fluids administered as Ringer's lactate (minimum of 20 mL/kg) at the discretion of the attending anesthesiologist. All incision sites were infiltrated with 0.25% bupivacaine, and CO2 insufflation pressure was limited to a maximum of 15 mmHg.

At the end of the procedure injections will be given by the surgeon through trocars intraperitoneally, then isoflurane will be discontinued and, the neuromuscular blockade will be antagonized by using neostigmine 0.05mg/kg plus atropine 0.01 mg/kg after assessment by nerve stimulator according to the train of four and will be administered to reverse the effect of rocuronium. then the trachea will be extubated, all patients will be transferred to the post-anesthesia unit (PACU). After completion of the surgical procedure, patients will be transferred to the post-anesthetic care unit (PACU), and the Modified Aldrete Score will be assessed and discharged after fulfilling an Aldrete score of ≥9.

To achieve blinding, the study drugs will be prepared in a ready-to-inject form by a separate anesthesiologist who is not involved in the study. This way, neither the patient nor the anesthesiologist administering the drug will be aware of the type of medication being used. The physician who will gather patient data is also unaware of the medications administered. During the first 24 hours After surgery, all patients will receive post-operative pain protocol (1 gm paracetamol IV every 8 hr.).

Pethidine 0.5 mg/kg diluted in 5 ml, titrated IV as rescue analgesia if VAS is greater than 3, or at any time the patient demands additional analgesia.

In the presence of nausea, with or without vomiting, granisetron 1 mg will be given intravenously and repeated if nausea persists (maximum dose of 3 mg per day).

Complications including postoperative nausea, vomiting, and other complications related to the drug used (e.g., toxicity,) will be recorded up to 24 hours after surgery.

The intensity of postoperative abdominal and shoulder pain will be measured on arrival in the recovery room and subsequently at time intervals of 2, 4, 6, 12, and 24 h using a 10-cm linear visual analog scale (VAS). The scale consisted of a horizontal line marked ''no pain' at one end and ''worst pain' at the other. Abdominal pain scores were measured at rest (supine), with activity (sitting up from supine), and with coughing. The time interval from extubation to the first administration of nalbuphine will be registered. The consumption of postoperative analgesics was recorded. Side effects (nausea, vomiting, sweating, dizziness, tinnitus, muscular twitches, and circumoral numbness), and recovery variables (return of bowel function, time interval to ambulation, resumption of liquid intake, and hospital discharge) will be assessed by the ward nurses at 2-h intervals. Patients were immediately given 1 mg intravenous granisetron and repeated if nausea persisted (maximum dose of 3 mg per day).

if they experience nausea or vomiting. Patients will be deemed ready for discharge from the hospital when they are afebrile, vital signs are stable, oral nutrition (liquid) was tolerated without discomfort, and bowel function has returned. Bowel recovery time was defined as the time from the end of anesthesia until the presence of good intestinal sound (estimated by the same surgeon) or the first passage of flatus.

Outcome measures:

* Primary outcome:

  > Post-operative pain severity by VAS (at 0 (the point of full recovery state at PACU), 6 hr., 12 hr., 18 hr., and 24 hr.) will be assessed.
* Secondary outcomes:

  * Cumulative postoperative opioid consumption (total amount of opioid consumption) in the first 24 hours postoperatively.
  * The onset of the first analgesic request. (Time of rescue analgesia).
  * Patient satisfaction after 1st postoperative day (four-point scale (1 =excellent, 2= good, 3= fair,4= poor)).
  * Incidence of postoperative nausea and vomiting.
  * Incidence of complications (LA toxicity,).
  * The hemodynamics of the patients (mean ABP, HR) will be measured at 0 hr., 6 hr., 12 hr., 18 hr., and 24 hr. after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status 1-2 scheduled for a Laparoscopic gynecological procedure.

Exclusion Criteria:

* History of allergy to the medications used in the study.
* Contraindication as local infection at the site of port insertion.
* Severe cardiac (NYHA ≥Ⅲ or pulmonary dysfunction (known COPD, previous thoracic surgeries, or recent pulmonary infection).
* Severe hepatic impairment (Child C) (INR≥2, Albumin≤2.5).
* Severe Renal dysfunction (creatinine clearance < 30).
* Neurologic, a psychiatric or mental disorder affecting the patient's ability to interpret VAS score.
* Body mass index (BMI) ≥ 40 or ≤ 18 kg/m2.
* Patients who were converted to open surgery.
* ASA Ⅲ-Ⅳ.
* Patient refusal.
* Emergency operations.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
effect on postoperative pain control | 24 hours after the procedure
  Assessment of postoperative pain severity by Visual analog score (VAS score) (at 0 (the point of full recovery state at PACU), 6 hr., 12 hr., 18 hr., and 24 hr. after the end of the procedure) will be assessed.

SECONDARY OUTCOMES:
Postoperative opioid consumption | 24 hours after the procedure
  Cumulative postoperative opioid consumption (total amount of opioid consumption) in the first 24 hours postoperatively.
The onset of the first analgesic request | Within 24 hours after the procedure
  The onset of the first analgesic request. (Time of rescue analgesia). we will document the time when the patient asks for rescue analgesia
Patient satisfaction | After 24 hours of the procedure
  Patient satisfaction after first postoperative day (four-point scale (1 =excellent, 2= good, 3= fair,4= poor)).
Incidence of postoperative side effects | Within 24 hours after the procedure
  Incidence of postoperative side effects like nausea and vomiting

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Memedov, C. et al. (2008) "Comparison of analgesic effects of intraperitoneal Lornoxicam and Ropivacaine administration in laparoscopic cholecystectomy.," Medical Journal of Trakya University [Preprint]. Available at: https://doi.org/10.5174/tutfd.2008.01046.2.
- [Background] Cunningham TK, Draper H, Bexhell H, Allgar V, Allen J, Mikl D, Phillips K. A double-blinded randomised controlled study to investigate the effect of intraperitoneal levobupivacaine on post laparoscopic pain. Facts Views Vis Obgyn. 2020 Oct 8;12(3):155-161. PMID 33123690
- [Background] Wei X, Yao X. The Impact of Intraperitoneal Levobupivacaine on Pain Relief After Laparoscopic Cholecystectomy: A Meta-analysis of Randomized Controlled Studies. Surg Laparosc Endosc Percutan Tech. 2020 Feb;30(1):1-6. doi: 10.1097/SLE.0000000000000742. PMID 31913214
- [Background] Elnabtity AM, Ibrahim M. Intraperitoneal dexmedetomidine as an adjuvant to bupivacaine for postoperative pain management in children undergoing laparoscopic appendectomy: A prospective randomized trial. Saudi J Anaesth. 2018 Jul-Sep;12(3):399-405. doi: 10.4103/sja.SJA_760_17. PMID 30100838
- [Background] Gago Martinez A, Escontrela Rodriguez B, Planas Roca A, Martinez Ruiz A. Intravenous Ibuprofen for Treatment of Post-Operative Pain: A Multicenter, Double Blind, Placebo-Controlled, Randomized Clinical Trial. PLoS One. 2016 May 6;11(5):e0154004. doi: 10.1371/journal.pone.0154004. eCollection 2016. PMID 27152748
- [Background] Kroll PB, Meadows L, Rock A, Pavliv L. A multicenter, randomized, double-blind, placebo-controlled trial of intravenous ibuprofen (i.v.-ibuprofen) in the management of postoperative pain following abdominal hysterectomy. Pain Pract. 2011 Jan-Feb;11(1):23-32. doi: 10.1111/j.1533-2500.2010.00402.x. PMID 20642488
- [Background] Moss JR, Watcha MF, Bendel LP, McCarthy DL, Witham SL, Glover CD. A multicenter, randomized, double-blind placebo-controlled, single dose trial of the safety and efficacy of intravenous ibuprofen for treatment of pain in pediatric patients undergoing tonsillectomy. Paediatr Anaesth. 2014 May;24(5):483-9. doi: 10.1111/pan.12381. Epub 2014 Mar 20. PMID 24646068
- [Background] Raof RA, El Metainy SA, Alia DA, Wahab MA. Dexmedetomidine decreases the required amount of bupivacaine for ultrasound-guided transversus abdominis plane block in pediatrics patients: a randomized study. J Clin Anesth. 2017 Feb;37:55-60. doi: 10.1016/j.jclinane.2016.10.041. Epub 2016 Dec 28. PMID 28235529